CLINICAL TRIAL: NCT05352282
Title: Comparative Study Between the Efficacy of The Serratus Anterior Plane Block and Lumbar Intrathecal Fentanyl Injection for Postoperative Analgesia After Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Nozahy, resident doctor at anesthesia and ICU department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Soh-Med-22_03_02
Record Dates: First submitted 2022-04-17; First posted 2022-04-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Patients Undergoing Modified Radical Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Procedure: Serratus Anterior Plane Block
- Group B (Active Comparator)
  Interventions: Procedure: Lumbar Intrathecal Fentanyl Injection

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block — SAPB will be done preoperative before induction of anesthesia under songraphic guidance and aseptic conditions with the patient in the lateral position, with the side of the surgical side up and the upper limb hanging over the patient's head. The ribs will be then counted, and when the 5th rib is identified, the high-frequency probe will be put over it, in the mid-axillary line in a sagittal plane. The ribs, pleura, overlying serratus muscle and latissimus dorsi muscle will be identified, and the needle will be advanced cephalic in-plane until the tip reaches the plane between the serratus anterior and latissimus dorsi. Afterward, 2 mL dextrose 5% will be injected; then, 30 mL of bupivacaine 0.25% will be injected in the plane between the serratus anterior and latissimus dorsi.
  Arms: Group A
Procedure: Lumbar Intrathecal Fentanyl Injection — Patients will receive 25 microgram intracthecal fentanyl immediately preoperative.
  Arms: Group B

SUMMARY:
Modiﬁed radical mastectomy (MRM) is one of the most common surgeries performed, and one that may be associated with signiﬁcant acute postoperative pain in breast surgery. Acute postoperative pain is an independent risk factor in the development of chronic post-mastectomy pain .

Various regional anesthetic procedures have been tried to provide better acute pain control and, consequently, less chronic pain. They can reduce perioperative opiates requirement and thereby decreasing their possible side effects. These regional procedures include local wound inﬁltration, lumbar intrathecal fentanyl injection, thoracic epidural, thoracic paravertebral block (PVB), and ultrasound (US)-guided interfascial plane blocks. Currently, Ultrasound (US)-guided interfascial plane blocks have been recommended as safe, easy, and reliable alternatives to the use of thoracic epidural and paravertebral blocks in providing analgesia for patients about to undergo breast surgery.

Serratus anterior plane block (SAPB) is one of the Ultrasound (US)-guided interfascial plane blocks, it blocks the intercostal nerves II-VI by injection above or below the serratus muscle in the mid-axillary line and spares the pectoral nerves.

We assumed that SAPB could safely provide a better analgesic proﬁle with an opioid-sparing effect than Intrathecal fentanyl. We will perform this study to evaluate this assumption.

ELIGIBILITY:
Inclusion Criteria:

* 50 patients with American Society of Anesthesiologists (ASA) grade I to II, 18 to 60 years of age scheduled for Modified Radical Mastectomy surgery

Exclusion Criteria:

* Patient refusal.
* Patient with significant neurological , psychiatric or neuromuscular disease
* Alcoholism .
* Drug abuse .
* Pregnancy or lactating women .
* Suspected Coagulopathy .
* Morbid obesity .
* Known allergy to study medications .
* Septicaemia and local infection at the block site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
analgesic effect of serratus anterior plane block and lumbar intrathecal fentanyl injection after modified radical mastectomy | 1 year
  compare the analgesic effect between serratus anterior plane block and lumbar intrathecal fentanyl injection by using visual analogue score (vas).
  -Postoperative pain will be assessed using visual analog score (VAS) [0-10]. 0 - 3 mild pain 4 - 6 moderate pain 7 - 10 severe pain 10 <unbearable pain)

SECONDARY OUTCOMES:
Hemodynamics effects of serratus anterior plane block and lumbar intrathecal fentanyl injection in patient undergoing modified radical mastectomy | 1 year
  compare between serratus anterior plane block and lumbar intrathecal fentanyl injection as regard, hemodynamics of patient undergoing modified radical mastectomy.
  -The heart rate (HR), noninvasive arterial systolic blood pressure (SBP), diastolic blood pressure (DBP) and peripheral oxygen saturation (SpO2) will be recorded at baseline, after induction and with skin incision and every 5 minutes intraoperative till the end of surgery. And postoperative at 30 min, 1, 2, 3, 6, 12 and 24 hours.
Intra venous analgesics consumption after serratus anterior plane block and lumbar intrathecal fentanyl injection in patient undergoing modified radical mastectomy | one year
  compare between serratus anterior plane block and lumbar intrathecal fentanyl injection in patient undergoing modified radical mastectomy as regard intra venous analgesics consumption.
  All patients will receive paracetamol (15mg/KG/dose) immediately postoperative and after 6 hours. Patients will be assessed every one hour in the first 6 hours then every 3 hours in the next 18 hours.
  Patients will receive ketorolac 30 mg if VAS 3-5 . If VAS>5 ,morphine 0.1mg/kg will be given then total ketorolac and morphine consumption in 24 hours will be calculated and compared between both groups .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amaya F, Hosokawa T, Okamoto A, Matsuda M, Yamaguchi Y, Yamakita S, Taguchi T, Sawa T. Can acute pain treatment reduce postsurgical comorbidity after breast cancer surgery? A literature review. Biomed Res Int. 2015;2015:641508. doi: 10.1155/2015/641508. Epub 2015 Oct 1. PMID 26495309
- [Background] Wang L, Guyatt GH, Kennedy SA, Romerosa B, Kwon HY, Kaushal A, Chang Y, Craigie S, de Almeida CPB, Couban RJ, Parascandalo SR, Izhar Z, Reid S, Khan JS, McGillion M, Busse JW. Predictors of persistent pain after breast cancer surgery: a systematic review and meta-analysis of observational studies. CMAJ. 2016 Oct 4;188(14):E352-E361. doi: 10.1503/cmaj.151276. Epub 2016 Jul 11. PMID 27402075
- [Background] Garg R, Bhan S, Vig S. Newer regional analgesia interventions (fascial plane blocks) for breast surgeries: Review of literature. Indian J Anaesth. 2018 Apr;62(4):254-262. doi: 10.4103/ija.IJA_46_18. PMID 29720750
- [Background] Garg R. Regional anaesthesia in breast cancer: Benefits beyond pain. Indian J Anaesth. 2017 May;61(5):369-372. doi: 10.4103/ija.IJA_292_17. No abstract available. PMID 28584344